CLINICAL TRIAL: NCT06484361
Title: Phase II Monocentric Study to Evaluate a Novel Approach for Staging Prostate Cancer Patients by Using a Fully Integrated Hybrid PET/MRI
Brief Title: PET/MRI to Stage Prostate Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Maria Picchio, Associate professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PETMR-Staging-PCa1
Record Dates: First submitted 2023-03-22; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; BAY 86-7548

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Dual tracer PET/MRI
  Interventions: Drug: 68Ga-PSMA; Drug: 68Ga-RM2

INTERVENTIONS:
Drug: 68Ga-PSMA — all patients will undergo PET/MRI with 68Ga-PSMA and 68Ga-RM2 prior to surgical intervention
Drug: 68Ga-RM2 — all patients will undergo PET/MRI with 68Ga-PSMA and 68Ga-RM2 prior to surgical intervention

SUMMARY:
The main goal of this phase II clinical trial is to define a novel approach of staging prostate cancer (PCa) patients by using a fully integrated positron emission tomography/ magnetic resonance imaging (PET/MRI) system with 68Ga-prostate specifica membrane antigen (PSMA) and 68Ga-RM2 (bombesin antagonist).

50 patients with biopsy proven PCa will be studied by PET/MRI with 68Ga-PSMA and with 68Ga-RM2 and then will undergo prostatectomy and pelvic lymphadenectomy.

DETAILED DESCRIPTION:
This is a prospective monocentric open study (Phase II study). The study will include 50 consecutive PCa patients who will be recruited in the first 36 months of the study. All clinical and pathological variables available at the time of PET/MRI will be recorded for each patient and all patients will take a blood sample before the first PET/MRI study. All patients will undergo 68Ga-PSMA and 68Ga-RM2 PET/MRI studies at San Raffaele Hospital in two different days (> 48 hours between the two studies) and within one month from each other.

Then, patients will undergo surgical intervention (prostatectomy and pelvic/retroperitoneal lymphadenectomy) and the surgically removed prostate will be fixated and processed. Ex-vivo 3T-MRI study will be performed on the processed specimen (prostate gland) and afterwards, the prostate will be examined by a dedicated pathologist. Spatial coregistration of in vivo, ex-vivo and histopathological images will be performed so that the annotation (dominant tumor lesion) made by the pathologist will be translated onto in vivo PET/MR images and semi-quantitative and radiomic features will be extracted from PET and mp-MRI images

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old
* Biopsy proven high-grade PCa referred to prostatectomy and pelvic/retroperitoneal lymphadenectomy.
* Willing to provide a signed informed consent

Exclusion Criteria:

* Age < 18 years-old
* Inability to complete the needed imaging examinations (i.e. severe claustrophobia)
* Any additional medical condition that may significantly interfere with study compliance
* All the contraindications for MRI study (i.e. pacemaker)
* Evidence of metastatic disease on conventional imaging contraindicating the surgical procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
To define the diagnostic accuracy of PET/MRI system with the novel tracers 68Ga-PSMA and 68Ga-RM2 for the localization of primary prostate cancer | baseline
  All patients will undergo PET/MRI with 68Ga-PSMA and 68Ga-RM2 and then imaging findings will be correlated to histopathological findings gathered after prostatectomy. Specifically, at the patient level, we will count the number of patients where the different imaging modalities identified at least one intraprostatic cancer lesion. At the lesion level, on the other hand, we will match the intraprostatic lesions identified at imaging with those detected at histopathological examination. Therefore, providing measures of sensitivity, specificity, PPV, NPV for each imaging modality investigated ( 68Ga-PSMA PET, 68Ga-RM2 PET and MRI) at the lesion level.

SECONDARY OUTCOMES:
To optimize PET/MRI with 68Ga-PSMA and 68Ga-RM2 protocol by using novel imaging technique to stage PCa patients. | baseline
  The image acquisition protocol will be adjusted to ensure high quality of the images and patient compliance (measured with the number of patients that will complete all study procedures)
To characterize the primary PCa phenotype in high-grade patients | baseline
  The correlation between Gleason Score and clinical data will be investigated with univariate and multivariate general linear models. Specifically, standardized uptake value (SUV)max and SUVmean of 68Ga-PSMA and 68Ga-DOTA-RM2, apparent diffusion coefficient (ADC)min and ADCmean, cellular markers in the peripheral blood, as well as radiomic features extracted from PET and mpMR images will be investigated.
To evaluate the stability and reproducibility of imaging features in mp-MRI with test-retest procedure. | baseline
  Mann-whitney test will be used to assess the difference in the radiomic features extracted two days apart from the same MRI sequences
To evaluate the diagnostic accuracy of PET/MRI with 68Ga-PSMA and 68Ga-RM2 to stage T, N and M parameters in PCa patients. | 24 months after baseline
  To assess PET/MRI diagnostic accuracy for PCa primary staging (N and M) with 68Ga-PSMA and 68Ga-RM2, PET/MRI whole body images will be evaluated by a Nuclear Medicine and Radiology expert physicians, being aware of the patients' medical history and results of other imaging modalities. Histological data will be used as gold standard for the evaluation of diagnostic accuracy when possible; conventional imaging/follow-up will be used for the confirmation of M parameter. In case of positive findings, a histologic confirmation will be obtained when technically feasible. In particular, pelvic and/or retroperitoneal lymph nodes dissection will be performed in all patients included in the study. A biopsy of the suspicious lesion would be considered when possible in patients with metastases located in other sites. The diagnostic accuracy for T, N and M parameters will be measured with sensitivity, specificity, PPV and NPV at the patient level.
To evaluate patient management based on PET/MRI studies. | 24 months
  It will be assessed in how many cases the PET/MRI studies affected the well-being patients, measured with survival analysis

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No